CLINICAL TRIAL: NCT04441840
Title: Immune and Recovery Modulating Impact of Probiotic Supplementation After Intense Resistance Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lindenwood University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB-19-161
Record Dates: First submitted 2020-06-12; First posted 2020-06-22 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Immune Markers; Complete Blood Count (CBC) With Platelet Differentials; Muscle Damage; Muscular Force Production; Countermovement Jump; Muscular Fatigue; Muscular Soreness

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The supplements were delivered in identical containers, each marked with a separate code marked on the outside of the supplement container. Once data collection, data entry, and statistical analysis was completely finished, the study code was broken.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Probiotic Culture (Active Comparator): Active culture of Bacillus Coagulans Dose: 1 x 10^9 colony forming units (CFU)
  Interventions: Dietary Supplement: Active Probiotic Culture
- Inactive Probiotic Culture (Active Comparator): Inactive culture of Bacillus Coagulans (GBI-30, 6086) - Marked as "StaImune" Dose: 1 x 10^9 colony forming units (CFU)
  Interventions: Dietary Supplement: Inactive Probiotic Culture

INTERVENTIONS:
Dietary Supplement: Active Probiotic Culture — Both conditions matched in appearance and serving size
  Arms: Active Probiotic Culture
Dietary Supplement: Inactive Probiotic Culture — Both conditions matched in appearance and serving size
  Other Names: StaImune
  Arms: Inactive Probiotic Culture

SUMMARY:
This study proposal seeks to examine the efficacy of probiotic supplementation at mitigating changes in immune function and recovery after completion of intense, stressful exercise while also allowing for a better understanding of its ability to promote recovery and maintenance of physical performance.

DETAILED DESCRIPTION:
Study Visit 1 - Familiarization:

During the familiarization visit, participants will first read and sign an IRB-approved informed consent document and complete a short form of the International Physical Activity Questionnaire (IPAQ). Participants will then have their height, weight, and body composition determined using Dual-Energy X-ray Absorptiometry (DEXA) (Hologic Discovery A). To standardize body composition assessment, participants will be required to observe an 8-hour fast and maintain a well-hydrated state. Each participant will provide a urine sample to confirm a hydrated stated through determination of a urine specific gravity values greater 1.020. Participants will then complete a peak oxygen consumption test (VO2Peak) using indirect calorimetry on a ParvoMedics TrueOne (Sandy, UT) metabolic cart interfaced to a motorized cycle ergometer (Lode Corival). The peak oxygen consumption test protocol will require each study participants to start at 100 watts before progressively increasing by 1 watt every two seconds. To determine whether maximal effort occurred a respiratory exchange ratio of >1.00 must be achieved.

Following the peak oxygen consumption assessment, participants will perform practice repetitions of all performance tests (force plate vertical jumps, isometric mid-thigh pulls, Biodex isometric and isokinetic knee extensor testing) as well as the exercises that will be performed during Visit 3 (leg press, hex bar deadlift, and drop jump).

Study Visit 2 - Pre-Supplementation Baseline Testing:

Study participants will be asked to complete a 24-hour food recall between each testing condition and will be asked to replicate their diet prior to this visit for all subsequent visits. Upon arrival, participants will first have their blood drawn from a forearm vein before completing a perceived soreness, pressure-pain threshold, and recovery assessment. Prior to testing, participants will complete the same standardized warm-up consisting of 5 minutes of light cycling, 10 body weight squats, 10 body weight walking lunges, 10 dynamic walking hamstring stretches (straight-leg march), and 10 dynamic walking quadriceps stretches. After the warm-up, participants will complete five countermovement jump squats on top of bilateral triaxial force plates (Hawkins Dynamics) interfaced to a personal computer to derive relevant force-time variables. Next, participants will complete two assessments of peak isometric force production. Using an electronic load cell with a 5,000-N capacity (Load Star load cells) connected to a computer, three 5-second maximal isometric mid-thigh pulls will be completed. Participants will then be outfitted on a Biodex isokinetic dynamometer where they will complete three maximal isometric knee extensions. Following the isometric knee extensor testing, participants will complete a 50-repetition test of concentric-only repetitions to assess changes in force production, torque, and rates of fatigue development. After the baseline performance testing, participants will have their leg press and hex bar deadlift one-repetition maximum (1RM) determined.

*Supplementation (14 days, described below) followed by exercise trial.*

Study Visit 3 (Post-Supplementation Testing, Exercise Trial):

Upon arrival, study participants will be asked to complete a 24-hour food recall and between each testing condition, study participants will be asked to replicate their diet. Upon arrival, participants will first have their blood drawn from a forearm vein before completing perceived soreness, pressure-pain threshold, and recovery assessments. Prior to testing, participants will complete the same standardized warm-up consisting of 5 minutes of light cycling, 10 body weight squats, 10 body weight walking lunges, 10 dynamic walking hamstring stretches (straight-leg march), and 10 dynamic walking quadriceps stretches. After the warm-up, participants will complete five countermovement jump squats on top of bilateral triaxial force plates (Hawkins Dynamics) interfaced to a personal computer to derive relevant force-time variables. Using an electronic load cell with a 5,000-N capacity (Load Star load cells) connected to a computer, three 5-second maximal isometric mid-thigh pulls will be completed. Participants will then be positioned on a Biodex isokinetic dynamometer where they will complete three maximal isometric knee extensions. Lastly, participants will complete a 50-repetition test of concentric-only repetitions to assess changes in force production, torque, and rates of fatigue development. Following the completion of these tests, participants will perform an exercise trial according to the methods described below. Following completion of the exercise trial, participants will undergo the previous testing battery (blood sample, perceived soreness, pressure-pain threshold assessment, recovery assessment, countermovement vertical jumps, isometric mid-thigh pulls, Biodex isometric and isokinetic testing) at five time points: immediately after exercise, 30 minutes post-exercise, 1 hour, 2 hours, and 5 hours post-exercise.

Study Visits 4 - 6: Post-Exercise Performance In an identical fashion, with the exception of 1RM assessment, study visits 4, 5, and 6 will be completed 24, 48, and 72 hours, respectively, after completion of the exercise bout. Briefly, study participants will return to the laboratory after an overnight fast (10 hours). Participants will bring in the completed 24-hour dietary recall, donate venous blood samples, assess their soreness, pressure-pain threshold, and recovery, complete the warm-up, perform five countermovement jumps, assess peak isometric force production, and complete a 50-repetition muscle fatigue test during each visit.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Free from any disorders or diseases as stated on health history form
* Between the ages of 18 - 55 years of age

Exclusion Criteria:

* Currently being treated for or are diagnosed with a cardiac, respiratory, circulatory, musculoskeletal, metabolic, obesity (defined as body mass index > 30 kg/m2 and body fat greater than 30%), immune, autoimmune, hematological, neurological or endocrinological disorder or disease unless the scenario is viewed to not be a contraindication by the clinical coordinator of the study protocol. Individuals who are currently prescribed a hypertensive or cholesterol-lowering medication will be allowed entry into the study with clearance from clinical coordinator or their personal physician.
* Female
* An individual who is less than 18 and greater than 55 years of age will be excluded.
* Participants younger than 18 are excluded due to necessity of parental consent.
* Participants greater than 55 years old lie outside of the target demographic for the current study.
* Considered to be sedentary, defined as getting less than 30 minutes of moderate intensity physical activity for most days of the week.
* Currently not resistance training at least 2 days per week for the past 30 days
* Currently smoking or have quit smoking within the past 6 months
* Currently taking a probiotic. Individuals who currently report as taking a probiotic will be allowed entry into study protocol if a wash-out period of 30 days is observed.)
* Currently consuming any form of dietary supplements that are viewed by study investigators to confound the outcomes of the study protocol (i.e., creatine, beta-alanine, essential amino acids, beta-hydroxy-beta-methylbutyrate (HMB), branched-chain amino acids, or any pre-workout that contain combinations of these ingredients). Individuals who currently report as taking any of these supplements will be allowed entry into study protocol if a wash-out period of 30 days is observed.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Immune Markers | Three weeks
  C-reactive protein [milligrams per liter (mg/L)]
Complete blood count | Three weeks
  White blood cell and platelet count [Thousand per microliter (Thousand/uL)]
Markers of muscle damage | Three weeks
  Creatine kinase [Units per liter (U/L)]
Force production assessment | Three weeks
  Maximal voluntary isometric contraction (knee extension) [pounds (lb)]
Force production assessment | Three weeks
  Isometric mid-thigh pull [pounds (lb)]
Countermovement Jump | Three weeks
  peak force [Newtons (N)]
Countermovement Jump | Three weeks
  eccentric force [Newtons (N)]
Countermovement Jump | Three weeks
  eccentric rate of force development [Newtons (N)]
Countermovement Jump | Three weeks
  reactive strength index
Dynamic muscular fatigue | Three weeks
  Biodex 50-repetition test [Percent fatigue rate]
Perceived soreness | Three weeks
  Soreness questionnaire (0 - 10) 0 is low, 10 is high
Perceived soreness | Three weeks
  pain-pressure threshold via algometer [Newtons (N)]
Immune Marker | Three weeks
  Interleukin-6, Tumor necrosis factor-alpha, Monocyte chemoattractant protein 1 [picograms per milliliter (pg/mL)]
Markers of muscle damage | Three weeks
  Myoglobin [nanogram per milliliter (ng/mL)].
Complete blood count (CBC) | Three weeks
  Red blood cell count [Millions per microliter (million/uL)]
Complete blood count (CBC) | Three weeks
  Hemoglobin and Mean corpuscular hemoglobin concentration (MCHC) [grams per deciliter (g/dL)]
Complete blood count (CBC) | Three weeks
  Hematocrit, neutrophils, lymphocytes, monocytes, eosinophils, basophils,Red cell distribution width (RDW) [Percentage (%)]
Complete blood count (CBC) | Three weeks
  Mean corpuscular volume (MCV) and Mean platelet volume (MPV) [Femtoliters (fL)]
Complete blood count (CBC) | Three weeks
  Mean corpuscular hemoglobin (MCH) [Picograms (pg)]
Complete blood count (CBC) | Three weeks
  Absolute neutrophils, absolute lymphocytes, absolute monocytes, absolute eosinophils, absolute basophils [cells per microliter (cells/uL)]

CONTACTS AND LOCATIONS:
Overall Officials: Chad Kerksick, PhD, Principal Investigator — Laboratory Director
Locations (1):
- Lindenwood University, Saint Charles, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
All approved unidentified study data inside the laboratory will be saved within a research repository bank for future research questions. Otherwise, participant data will be destroyed after three years of study completion to maintain Institutional Review Board (IRB) compliance